CLINICAL TRIAL: NCT06848985
Title: Impact of Combined Aerobic and Resistance Exercise on Autonomic Function and Cardiopulmonary Endurance in Obese College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital University of Physical Education and Sports, China (Other)
Responsible Party: Principal Investigator, Bai Shuang, Doctor, Beijing Sport University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.155223005
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Obese College Students; Aerobic Exercise Combined with Resistance Exercise
Keywords: Aerobic exercise combined with resistance exercises; Cardiorespiratory endurance; Autonomic function; Obese college students

STUDY DESIGN:
Intervention Model Description: Obese college students aged 18-22 were recruited from a university in Beijing to participate in a public elective course on exercise for weight loss and slimming at the Capital University of Physical Education and Sport (CUPES). Ultimately, 60 students who met these criteria were selected for the study, divided into an experimental group of 30 and a control group of 30. The study primarily utilized a combined exercise regimen of aerobic and resistance exercises, conducted three times a week over a period of 16 weeks. The control group maintained their normal physical activity levels without any additional intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): 30 participants underwent a 16-week program of aerobic (60%-70% HRmax for 40 minutes) and resistance exercises (65%-70% RM for 30 minutes).
  Interventions: Behavioral: Aerobic combined with Resistance exercise
- Control Group (No Intervention): 30 participants maintained normal physical activity without additional interventions.

INTERVENTIONS:
Behavioral: Aerobic combined with Resistance exercise — Participants are required to perform aerobic and resistance exercises. Aerobic exercises included the use of treadmills and elliptical machines, with intensity maintained at 60%-70% of the maximum heart rate (calculated as 220 minus age), for a total of 40 minutes per session (5 minutes of warm-up, 30 minutes of main exercise, and 5 minutes of cool-down). Heart rate monitors were used to ensure the intensity was maintained; resistance exercises involved gym equipment and bodyweight exercises, including the use of a pec deck machine, lat pull-downs, chest presses, bicep curls, tricep extensions, leg curls, and leg presses. The intensity of resistance exercises was set at about 65%-70% of one repetition maximum (1RM), with each session consisting of three sets of 6-8 repetitions and lasting for 30 minutes.
  Arms: Experimental Group

SUMMARY:
This study explores the potential link between aerobic exercise combined with resistance training and improvements in cardiopulmonary function in obese individuals, focusing particularly on the influence of autonomic nerve function. By examining the effects of combined exercise on obese college students, this research aims to elucidate the critical role that autonomic nerve function improvement plays in enhancing cardiopulmonary function in this demographic.

The study primarily utilized a combined exercise regimen of aerobic and resistance exercises, conducted three times a week over a period of 16 weeks. One session was held during class hours, with the remaining two sessions scheduled during free time in the university gym. Aerobic exercises included the use of treadmills and elliptical machines, with intensity maintained at 60%-70% of the maximum heart rate (calculated as 220 minus age), for a total of 40 minutes per session (5 minutes of warm-up, 30 minutes of main exercise, and 5 minutes of cool-down). Heart rate monitors were used to ensure the intensity was maintained; resistance exercises involved gym equipment and bodyweight exercises, including the use of a pec deck machine, lat pull-downs, chest presses, bicep curls, tricep extensions, leg curls, and leg presses. The intensity of resistance exercises was set at about 65%-70% of one repetition maximum (1RM), with each session consisting of three sets of 6-8 repetitions and lasting for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Obese college students aged 18-22 were recruited from a university in Beijing to participate in a public elective course on exercise for weight loss and slimming at the Capital University of Physical Education and Sport (CUPES). The inclusion criteria included a BMI of ≥28 kg/m^2, no history of chronic diseases such as cardiovascular or metabolic diseases, no psychiatric conditions (e.g., depression, anxiety disorder, obsessive-compulsive disorder), and no physical disabilities or movement disorders (such as bone and joint diseases).

Exclusion Criteria:

* The exclusion criteria include individuals with diseases that may affect training (such as cardiovascular diseases, respiratory diseases, and musculoskeletal disorders), as well as those diagnosed with mental disorders (such as depression, anxiety, obsessive-compulsive disorder, etc.).

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-09-02 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
Autonomic function | From enrollment to the end of treatment at 16 weeks
  Autonomic function was assessed using the Pushikang FLY-2 autonomic physiological monitor. Participants were required to abstain from caffeinated and alcoholic beverages for 12 hours and from strenuous physical activity for 48 hours prior to the test. The testing was conducted between 8:00 a.m. and 11:00 a.m. in a controlled environment with temperatures maintained at 22-24°C. The test duration was 5 minutes, during which participants sat quietly and refrained from speaking. Autonomic nerve function parameters were recorded using finger photoplethysmography to measure pulse wave changes in a resting state. Data was processed using Beijing Fourier's autonomic nerve response analysis software (ANS-1, V6.6). Time-domain analysis focused on the mean interval between heartbeats to reflect sympathetic/vagal modulation, and the variance of these intervals indicated the overall variability of cardiac function, providing critical prognostic information.
Cardiorespiratory endurance | From enrollment to the end of treatment at 16 weeks
  Cardiopulmonary function was evaluated using the cardiopulmonary exercise test (CPET, Schiller) on a Rehab-B exercise treadmill. To ensure test accuracy, participants were instructed to refrain from physical activity on the day prior to the test and to avoid alcohol, caffeinated beverages, and food for 8 hours before testing and during the first 3 hours of the test day. The exercise commenced with a 3-minute rest followed by a gradual load phase, allowing participants to reach voluntary fatigue within 8 to 12 minutes, and then continue at maximum tolerance for an additional 3 minutes. The exercise protocol followed the Bruce protocol, with incremental loads adjusted for gender: 25 W/min for males and 15 W/min for females.

SECONDARY OUTCOMES:
The Functional Movement Screen (FMS) score | From enrollment to the end of treatment at 16 weeks
  The Functional Movement Screening (FMS) is a standardized tool used to assess the functional motor abilities of individuals. It consists of seven tests (squatting, stepping, lunging, reaching, leg raising, push-up, and rotary stability) that balance flexibility and stability, allowing medical and fitness professionals to identify problems such as weakness, imbalance, asymmetry, and movement limitations. In the FMS, each action is scored from 0 to 3: a score of 3 indicates the individual can perform the movement standardly and stably without compensation; a score of 2 signifies that the movement can be completed, albeit with some instability or compensatory behavior; a score of 1 indicates an inability to perform the movement according to the standards. Research has shown that lower FMS scores correlate with a higher risk of injury. Typically, a threshold score of 14 is used, with individuals scoring below this level considered at greater risk of injury.
Body composition | From enrollment to the end of treatment at 16 weeks
  Body composition was assessed using the InBody760 (Ver. LookinBody120.4.0.0.7) bioelectrical impedance analyzer. Measurements were taken in the early morning, with subjects fasting and in a controlled temperature environment (22-24℃), providing immediate readings of body mass index (BMI), body fat percentage, waist-to-hip ratio, visceral fat area.

CONTACTS AND LOCATIONS:
Locations (1):
- Capital University Of Physical Education And Sports, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code